CLINICAL TRIAL: NCT01524276
Title: Medtronic Product Surveillance Registry
Brief Title: Product Surveillance Registry
Acronym: PSR
Status: Recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PSR
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Rhythm Disorders; Urological Disorders; Neurological Disorders; Cardiovascular Disorders; Digestive Disorders; Intracranial Aneurysm; Mechanical Circulatory Support; Respiratory Therapy; Aortic, Peripheral Vascular and Venous Disorders; Minimally Invasive Surgical Procedures; Diagnostic Techniques and Procedures; Surgical Procedures, Operative; Renal Insufficiency; Neurovascular; Coronary Artery Disease; Ear, Nose and Throat Disorder
MeSH Terms: conditions — Urologic Diseases; Nervous System Diseases; Cardiovascular Diseases; Digestive System Diseases; Intracranial Aneurysm; Renal Insufficiency; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Registry is to provide continuing evaluation and periodic reporting of safety and effectiveness of Medtronic market-released products. The Registry data is intended to benefit and support interests of patients, hospitals, clinicians, regulatory bodies, payers, and industry by streamlining the clinical surveillance process and facilitating leading edge performance assessment via the least burdensome approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible Medtronic product
* Patient within enrollment window relative to therapy initiation or meets criteria for retrospective enrollment

Exclusion Criteria:

* Patient who is, or will be, inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with Medtronic qualifying therapy product.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2012-01; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Effectiveness of Market Released products | Every 6-12 months (Therapy-dependent)

CONTACTS AND LOCATIONS:
Locations (387):
- United States (131):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Aliso Viejo, California
  - Chula Vista, California
  - Colton, California
  - La Jolla, California
  - Los Angeles, California
  - Napa, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Darien, Connecticut
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Davie, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Panama City, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Weston, Florida
  - Gainesville, Georgia
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Hyattsville, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Holyoke, Massachusetts
  - Ann Arbor, Michigan
  - Bay City, Michigan
  - Lansing, Michigan
  - Rochester Hills, Michigan
  - Ypsilanti, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Camden, New Jersey
  - Marlton, New Jersey
  - Morristown, New Jersey
  - Ocean Township, New Jersey
  - Teaneck, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Bay Shore, New York
  - Huntington, New York
  - Manhasset, New York
  - Mount Kisco, New York
  - New Hyde Park, New York
  - New York, New York
  - Poughkeepsie, New York
  - Riverhead, New York
  - Roslyn, New York
  - Staten Island, New York
  - Stony Brook, New York
  - Utica, New York
  - Chapel Hill, North Carolina
  - Charleston, North Carolina
  - Durham, North Carolina
  - Eatonton, North Carolina
  - Pinehurst, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Mount Orab, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Mechanicsburg, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Spartanburg, South Carolina
  - Sioux Falls, South Dakota
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Kyle, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Fredericksburg, Virginia
  - Bremerton, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Buenos Aires, Argentina
- Australia (4):
  - Westmead, New South Wales
  - Chermside
  - Murdoch
  - Southport
- Austria (2):
  - Innsbruck
  - Linz
- Belgium (10):
  - Aalst
  - Bruges
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Leuven
  - Liège
  - Roeselare
  - Sint-Niklaas
- São Paulo, Brazil
- Canada (5):
  - Calgary, Alberta
  - Kingston, Ontario
  - Montreal, Quebec
  - Québec
  - Toronto
- China (11):
  - Chengdu, Sichuan
  - Beijing
  - Chengdu
  - Dalian
  - Guangzhou
  - Hangzhou
  - Harbin
  - Kunming
  - Nanchang
  - Shanghai
  - Suzhou
- Colombia (4):
  - Cartagena
  - Medellín
  - Pereira
  - Rionegro
- Prague, Czechia
- Denmark (4):
  - Copenhagen
  - Hellerup
  - Hillerød
  - Odense
- Finland (2):
  - Helsinki
  - Tampere
- France (24):
  - Avignon
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Caen
  - Chambray
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - La Rochelle
  - La Tronche
  - Lille
  - Marseille
  - Montpellier
  - Nantes
  - Ollioules
  - Paris
  - Pessac
  - Pringy
  - Rennes
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Villeurbanne
- Germany (24):
  - Aachen
  - Arnsberg
  - Bad Oeynhausen
  - Berlin
  - Bochum
  - Bremen
  - Cologne
  - Düsseldorf
  - Freiburg im Breisgau
  - Hagen
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Jena
  - Karlsruhe
  - Leipzig
  - Lübeck
  - München
  - Münster
  - Stuttgart
  - Tübingen
  - Ulm
  - Wiesbaden
- Greece (3):
  - Athens
  - Marousi
  - Thessaloniki
- Hong Kong, Hong Kong
- Budapest, Hungary
- India (8):
  - Jaipur, Rajasthan
  - Hyderabad, Telangana
  - Bangalore
  - Bengaluru
  - Chennai
  - Gūrgaon
  - Kochi
  - New Delhi
- Galway, Ireland
- Israel (4):
  - Ashkelon
  - Beersheba
  - Jerusalem
  - Ramat Gan
- Italy (18):
  - Acquaviva delle Fonti
  - Ancona
  - Bari
  - Bologna
  - Brescia
  - Caserta
  - Castrovillari
  - Cotignola
  - Lecce
  - Milan
  - Modena
  - Monza
  - Palermo
  - Pisa
  - Roma
  - Rome
  - Taranto
  - Udine
- Japan (34):
  - Sakai, Osaka
  - Ageo, Saitama
  - Hidaka, Saitama
  - Koshigaya, Saitama
  - Tokyo, Tachikawa
  - Bunkyō-Ku, Tokyo
  - Minato-Ku, Tokyo
  - Yonago, Tottori
  - Chiba
  - Fukui
  - Fukuoka
  - Gifu
  - Hirosaki
  - Hiroshima
  - Kagoshima
  - Kamakura
  - Kawasaki
  - Kitakyushu
  - Kofu
  - Kumamoto
  - Kyoto
  - Mitaka
  - Nagoya
  - Niigata
  - Okayama
  - Ōsaka-sayama
  - Sapporo
  - Shinagawa-Ku
  - Shizuoka
  - Suita
  - Tokyo
  - Toyoake
  - Urasoe
  - Yokohama
- Kuwait City, Kuwait
- Kuala Lumpur, Malaysia
- Mexico City, Mexico
- Netherlands (12):
  - Amsterdam
  - Doetinchem
  - Eindhoven
  - Enschede
  - Groningen
  - Heerlen
  - Hengelo
  - Leiden
  - Maastricht
  - Nieuwegein
  - Rotterdam
  - The Hague
- Christchurch, New Zealand
- Norway (3):
  - Bergen
  - Lorenskog
  - Trondheim
- Panama City, Panama
- Poland (3):
  - Poznan
  - Warsaw
  - Zabrze
- Portugal (5):
  - Carnaxide
  - Creixomil
  - Lisbon
  - Porto
  - Santarém
- Puerto Rico (2):
  - Aibonito
  - Rio Piedras
- Saudi Arabia (2):
  - Jeddah
  - Riyadh
- Belgrade, Serbia
- Bratislava, Slovakia
- South Korea (14):
  - Yangsan, Gyeongsangnam-do
  - Busan
  - Changwon
  - Cheongju-si
  - Daegu
  - Daejeon
  - Gangneung
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeonju
  - Seongnam-si
  - Seoul
  - Suwon
- Spain (16):
  - A Coruña
  - Córdoba
  - Elche
  - Girona
  - Granada
  - L'Hospitalet de Llobregat
  - Madrid
  - Málaga
  - Palma de Mallorca
  - Salamanca
  - Santa Cruz de Tenerife
  - Santiago de Compostela
  - Toledo
  - Valencia
  - Valladolid
  - Vitoria-Gasteiz
- Sweden (3):
  - Gothenburg
  - Lund
  - Skövde
- Switzerland (8):
  - Basel
  - Bern
  - Fribourg
  - Geneva
  - Lausanne
  - Lugano
  - Morges
  - Zurich
- Taichung, Taiwan
- United Kingdom (17):
  - Barnstaple
  - Birmingham
  - Blackpool
  - Bristol
  - Chelmsford
  - Glasgow
  - Harrow
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Middlesbrough
  - Newcastle upon Tyne
  - Northampton
  - Sheffield
  - Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goya M, Park SJ, Ando K, Holbrook R, Iskandar R, Jacobsen L, Mozingo JD, Joung B; SPARK Registry Investigators. Safety and efficacy of an intrinsic antitachycardia pacing algorithm in patients from Japan and South Korea: results from a cardiac device registry in the Asia Pacific region. J Med Econ. 2025 Dec;28(1):1307-1318. doi: 10.1080/13696998.2025.2543213. Epub 2025 Aug 13. PMID 40758483
- [Derived] Patel D, Rao A, Friedman PA, Deshmukh AJ, Lande J, Murphy JA, Brown ML, Lexcen DR, Wilkoff BL. New atrial arrhythmia occurrence in single chamber implantable cardioverter defibrillator patients: A real-world investigation. J Cardiovasc Electrophysiol. 2023 Feb;34(2):438-444. doi: 10.1111/jce.15790. Epub 2022 Dec 30. PMID 36579406
- [Derived] Qin D, Filippaios A, Murphy J, Berg M, Lampert R, Schloss EJ, Noone M, Mela T. Short- and Long-Term Risk of Lead Dislodgement Events: Real-World Experience From Product Surveillance Registry. Circ Arrhythm Electrophysiol. 2022 Aug;15(8):e011029. doi: 10.1161/CIRCEP.122.011029. Epub 2022 Aug 4. PMID 35925831
- [Derived] Garg A, Koneru JN, Fagan DH, Stromberg K, Padala SK, El-Chami MF, Roberts PR, Piccini JP, Cheng A, Ellenbogen KA. Morbidity and mortality in patients precluded for transvenous pacemaker implantation: Experience with a leadless pacemaker. Heart Rhythm. 2020 Dec;17(12):2056-2063. doi: 10.1016/j.hrthm.2020.07.035. Epub 2020 Aug 4. PMID 32763431
- [Derived] Singh JP, Cha YM, Lunati M, Chung ES, Li S, Smeets P, O'Donnell D. Real-world behavior of CRT pacing using the AdaptivCRT algorithm on patient outcomes: Effect on mortality and atrial fibrillation incidence. J Cardiovasc Electrophysiol. 2020 Apr;31(4):825-833. doi: 10.1111/jce.14376. Epub 2020 Feb 28. PMID 32009263
- [Derived] Stearns LM, Abd-Elsayed A, Perruchoud C, Spencer R, Hammond K, Stromberg K, Weaver T. Intrathecal Drug Delivery Systems for Cancer Pain: An Analysis of a Prospective, Multicenter Product Surveillance Registry. Anesth Analg. 2020 Feb;130(2):289-297. doi: 10.1213/ANE.0000000000004425. PMID 31567325